CLINICAL TRIAL: NCT00397254
Title: An Observer-Blind, Randomized, Parallel-Group Study to Compare the Efficacy of Two Rizatriptan Prescribing Portions for the Treatment of Migraine
Brief Title: Two Rizatriptan Prescribing Portions for Treatment of Migraine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Clinvest (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Roger K. Cady, MD, Clinvest
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 078-00
Record Dates: First submitted 2006-11-07; First posted 2006-11-09 (Estimated); Results first posted 2009-09-22 (Estimated); Last update posted 2010-06-08 (Estimated); Status verified 2009-09

CONDITIONS: Migraine
Keywords: Migraine; rizatriptan
MeSH Terms: conditions — Migraine Disorders | interventions — rizatriptan

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clinical Limit (Active Comparator): Eligible patients were randomized to one of two treatment regimens in a 1:1 ratio. Those randomized to receive a "clinical limit" of study medication received Rizatriptan 10mg ODT: 27 tablets per month.
  Interventions: Drug: rizatriptan
- Formulary Limit (Active Comparator): Eligible patients were randomized to one of two treatment regimens in a 1:1 ratio. Those randomized to receive a "formulary limit" of study medication received Rizatriptan 10mg ODT: 9 tablets per month.
  Interventions: Drug: rizatriptan

INTERVENTIONS:
Drug: rizatriptan — 10mg ODT 27 tablets
  Other Names: Maxalt
  Arms: Clinical Limit
Drug: rizatriptan — 10mg ODT 9 tablets
  Other Names: Maxalt
  Arms: Formulary Limit

SUMMARY:
The primary objective of this study is to evaluate a clinical limit (CL) of rizatriptan (9 rizatriptan 10mg Orally Disintegrating Tablet (ODT) per month) versus (vs.) a formulary limit (FL) of rizatriptan (27 rizatriptan 10mg ODT per month) as measured by the number of days of migraine per month.

DETAILED DESCRIPTION:
A common clinical perception exists that less effective treatment of attacks increases the burden of disease across attacks in the form of increased attack frequency, severity, duration, and/or treatability. If this perception is true, more effective treatment decreases the burden of disease across attacks. There are multiple barriers to effective treatment. The triptan class of migraine medications is frequently dispensed in the context of health benefit plan formulary limitations. Because of limited supply, medications must be used very cautiously. Patients may hoard medication in reaction to fear of running out. Overly cautious use and hoarding may lead to greater disease burden.

The purpose of this study is to compare the effect of two allocations of rizatriptan - a more limited allocation ("Formulary Limit") vs. a less limited allocation ("Clinical Limit") on disease burden.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age
* Patient has at least a 1-year history of migraine with or without aura by International Headache Society (IHS) criteria 1.1 and 1.2
* Patient typically has 3-8 migraine attacks/month
* Patient has less than 10 headache days/month with no evidence of IHS 8.2 Medication Overuse Headache
* Patient receives their triptan medication under a pre-determined prescribing allocation ranging from 6-12 tablets per month for the last 3 months preceding Visit 1.
* Patient and investigator agree that multiple doses of rizatriptan described in the package circular are appropriate for non-responsive or recurring headache.
* Patient uses a triptan as mainstay of acute therapy at Visit 1.
* Patient of childbearing potential agrees to use adequate contraception during the study. Adequate methods of contraception are to be determined by the investigator and should be consistent with contraceptive care administered in the regular clinical use of rizatriptan outside the study.
* Patient understands study procedures, alternative treatments available, and risks involved with the study, and voluntarily agrees to participate by giving written informed consent.

Exclusion Criteria:

* Patient has headache disorders beyond migraine or episodic tension-type headache IHS 2.1
* Patient is receiving prophylactic therapy for migraine
* Patient is currently taking:

Daily or nearly daily (typically >3 days out of 7 days) use of non-steroidal anti-inflammatory drugs (NSAIDs), COX-2 inhibitors, or other analgesics. Aspirin less than or equal to 325mg daily is allowed for cardioprotection.

Monoamine oxidase inhibitors (MAOIs) Propranolol Patient taking either an MAOI ro propranolol may be enrolled in the study, if in the clinical judgement of the investigator, either of these medications can be discontinued 2 weeks prior to study entry. Otherwise the use of MAOIs and propranolol are prohibited during the study.

* Patient has basilar or hemiplegic migraine headache.
* Patient has history or clinical evidence of ischemic heart disease (e.g., angina pectoris of any type, history of myocardial infarction or documented silent ischemia) or symptoms or finding consistent with ischemic heart disease, coronary artery vasospasm (including Prinzmetal's variant angina), or other significant underlying cardiovascular disease.
* Patient has uncontrolled hypertension.
* Patient has either demonstrated hypersensitivity to or experienced a serious adverse event in response to rizatriptan or any of its inactive ingredients.
* Patient is pregnant or a nursing mother.
* Patient has a history (within 1 year) or current evidence of drug or alcohol abuse.
* Patient has received treatment with an investigational device or compound within 30 days of the study (Visit 1).
* Patient had clinical evidence of significant pulmonary, renal, hepatic, endocrine, neurologic (apart from migraine), psychiatric or any other condition that, in the opinion of the investigator may confound the results of the study, pose an additional risk, or interfere with optimal participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2006-12; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger K Cady, MD, Principal Investigator — Clinvest
Locations (10):
- United States (10):
  - Brian Koffman, MD, Diamond Bar, California
  - San Francisco Clinical Research Center, San Francisco, California
  - Physician Associates, Oviedo, Florida
  - Dr. B. Abraham, PC, Snellville, Georgia
  - Dhiren Shah, MD, Prince Frederick, Maryland
  - Westside Family Medical Center, Kalamazoo, Michigan
  - Clinvest, Springfield, Missouri
  - Mercy Health Research / Ryan Headache Center, St Louis, Missouri
  - PharmQuest, Greensboro, North Carolina
  - Thomas Jefferson University Hospital Jefferson Headache Center, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Brandes JL, Visser WH, Farmer MV, Schuhl AL, Malbecq W, Vrijens F, Lines CR, Reines SA; Protocol 125 study group. Montelukast for migraine prophylaxis: a randomized, double-blind, placebo-controlled study. Headache. 2004 Jun;44(6):581-6. doi: 10.1111/j.1526-4610.2004.446006.x. PMID 15186302
- [Derived] Cady RK, Goldstein J, Silberstein S, Juhasz M, Ramsey K, Rodgers A, Hustad CM, Ho T. Expanding access to triptans: assessment of clinical outcome. Headache. 2009 Nov-Dec;49(10):1402-13. doi: 10.1111/j.1526-4610.2009.01532.x. Epub 2009 Oct 8. PMID 19817885

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3-month Baseline Period occurred prior to randomization to Clinical Limit or Formulary Limit groups. 42 subjects discontinued from total enrollment of 197: (2) Adverse Event (AE), (10) Lost to Follow Up (LFU), (11) Withdrew consent, (1) Pregnancy, (16) Failed to meet Inclusion/Exclusion at Visit 4 Randomization, (2) Other
Groups:
- Rizatriptan 27 Tablets - Clinical Limit: Eligible patients were randomized to one of two treatment regimens in a 1:1 ratio. Those randomized to receive a "clinical limit" of study medication received Rizatriptan 10mg orally disintegrating tablet (ODT): 27 tablets per month.
- Rizatriptan 9 Tablets - Formulary Limit: Eligible patients were randomized to one of two treatment regimens in a 1:1 ratio. Those randomized to receive a "formulary limit" of study medication received Rizatriptan 10mg orally disintegrating tablet (ODT): 9 tablets per month.
Period: Overall Study
Arm/Group | Rizatriptan 27 Tablets - Clinical Limit | Rizatriptan 9 Tablets - Formulary Limit
Started | 79 | 76
Completed | 77 | 74
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Baseline Period - Rizatriptan 9 Tablets: Prior to randomization at Visit 2 (to rizatriptan 9 tablets or rizatriptan 27 tablets), all subjects in Baseline were provided with 9 tablets of rizatriptan.
Arm/Group | Baseline Period - Rizatriptan 9 Tablets
Number analyzed (Participants) | 197
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 197
  >=65 years | 0
Age Continuous [Mean (Full Range); unit: years] | 42 [18 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173
  Male | 24
Region of Enrollment [Number; unit: participants]
  United States | 197

OUTCOME MEASURES:

1. Primary Outcome: Number of Days With Migraine
Time Frame: 6 months
Population: 197 enrolled in Baseline(BL). Analysis of BL Characteristics on 197. 42 discontinued (2 Adverse Event(AE),10 Lost to followup(LFU),11 Withdrew consent,1 Pregnant,16 Failed randomization criteria,2 Other). 155 randomized. 4/155 LFU. 151 in analysis(77 Clinical Limit/74 Formulary Limit). 143 completed all visits(74 Clinical Limit/69 Formulary Limit).
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Rizatriptan 27 Tablets - Clinical Limit | Rizatriptan 9 Tablets - Formulary Limit
Number analyzed (Participants) | 77 | 74
Days | 2.666 (1.297) | 2.738 (1.313)

2. Secondary Outcome: Number of Migraine Attacks
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Migraine attacks
Arm/Group | Rizatriptan 27 Tablets - Clinical Limit | Rizatriptan 9 Tablets - Formulary Limit
Number analyzed (Participants) | 77 | 74
Migraine attacks | 4.855 (2.093) | 4.399 (1.548)

3. Secondary Outcome: Percentage of Responders
Description: Percentage of Responders (50% decrease in attack frequency) of Formulary Limit Group versus Percentage of Responders (50% decrease in attack frequency) in Clinical Limit Group
Time Frame: 6 months
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Rizatriptan 27 Tablets - Clinical Limit | Rizatriptan 9 Tablets - Formulary Limit
Number analyzed (Participants) | 77 | 74
Percentage of Participants | 7.79 | 2.70

4. Secondary Outcome: Average Attack Duration
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Rizatriptan 27 Tablets - Clinical Limit | Rizatriptan 9 Tablets - Formulary Limit
Number analyzed (Participants) | 77 | 74
Hours | 11.569 (8.188) | 12.930 (9.192)

5. Secondary Outcome: Headache Severity of All Attacks
Description: 4-Point Headache Severity Scale (0 = No Pain / 1 = Mild Pain / 2 = Moderate Pain / 3 = Severe Pain)
Time Frame: 6 months
Population: as for outcome 1
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Rizatriptan 27 Tablets - Clinical Limit | Rizatriptan 9 Tablets - Formulary Limit
Number analyzed (Participants) | 77 | 74
Units on a scale | 1.50 [1.00 to 2.76] | 1.59 [1.00 to 3.00]

6. Secondary Outcome: Percentage of Attacks With Symptom Elimination at 2 Hours
Description: Percentage of attacks with elimination of all associated symptoms at 2 hours post-treatment in Formulary Limit Group versus percentage of attacks with elimination of all associated symptoms at 2 hours post-treatment in Clinical Limit Group
Time Frame: 6 months
Population: as for outcome 1
Measure: Number; unit: Percentage of attacks
Arm/Group | Rizatriptan 27 Tablets - Clinical Limit | Rizatriptan 9 Tablets - Formulary Limit
Number analyzed (Participants) | 77 | 74
Percentage of attacks | 58.35 | 56.60

7. Secondary Outcome: Percentage of Attacks With Return to Normal Ability to Perform Activities at 2 Hours Post-dose
Description: Percentage of attacks with mild, moderate or severely impaired ability to perform activities pre-treatment with return to normal function at 2 hours post-dose in Formulary Limit Group versus Clinical Limit Group
Time Frame: 6 months
Population: as for outcome 1
Measure: Number; unit: Percentage of attacks
Arm/Group | Rizatriptan 27 Tablets - Clinical Limit | Rizatriptan 9 Tablets - Formulary Limit
Number analyzed (Participants) | 77 | 74
Percentage of attacks | 50.74 | 48.67

8. Secondary Outcome: Adverse Experiences
Description: Participants with one or more Adverse Experiences (AEs) in Formulary Limit Group versus Clinical Limit Group collected from time patient provided informed consent until return at Visit 7 or through 14 days post-dosing of the last dose of study medication if serious adverse experience. Defined as any unfavorable and unintended change in structure, function, or chemistry of the body temporally associated with use of provided product whether or not considered related to use of the product. Includes any worsening of a preexisting condition temporally associated with use of provided product.
Time Frame: 6 months
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Rizatriptan 27 Tablets - Clinical Limit | Rizatriptan 9 Tablets - Formulary Limit
Number analyzed (Participants) | 77 | 74
Participants | 18 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator is free to publish results of it's part of the study in collaboration with the other investigators subsequent to the multicenter publication issued by Clinvest. Principal Investigator (PI) may publish results of it's data with copy of any manuscript for review to Clinvest 60 days prior to submission for publication.